CLINICAL TRIAL: NCT04145336
Title: 7 cm vs. 5 cm Pancreatic Stents for the Prevention of Post-ERCP Pancreatitis in High-risk Patients: a Multicentre, Single-blinded, Randomised Controlled Trial
Brief Title: 7 cm vs. 5 cm Pancreatic Stents for the Prevention of Post-ERCP Pancreatitis in High-risk Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY20191010-2
Record Dates: First submitted 2019-10-18; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: ERCP; PEP; Post-ERCP pancreatitis; Pancreatic duct stent
MeSH Terms: interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5cm PDS group (Active Comparator): All patients in this group receive 5cm 5-Fr PDS.
  Interventions: Device: 5cm 5-Fr PDS; Drug: Indomethacin
- 7cm PDS group (Experimental): All patients in this group receive 7cm 5-Fr PDS.
  Interventions: Device: 7cm 5-Fr PDS; Drug: Indomethacin

INTERVENTIONS:
Device: 5cm 5-Fr PDS — High-risk patients receive 5cm 5-Fr PDS
  Arms: 5cm PDS group
Device: 7cm 5-Fr PDS — High-risk patients receive 7cm 5-Fr PDS
  Arms: 7cm PDS group
Drug: Indomethacin — All patients without contraindications should be administrated with rectal indomethacin within 30 min before ERCP.

SUMMARY:
Acute pancreatitis is the most common complication of endoscopic retrograde cholangiopancreatography (ERCP). The incidence of post-ERCP pancreatitis (PEP) is estimated to be 10% to 15% in high-risk patients. Current guidelines recommend using pancreatic duct stent (PDS) for PEP prevention in high-risk patients, but it is not clear whether stent length will affect the effect of PEP prevention. The longer PDS will remain in the pancreatic duct for a longer period of time, thereby ensuring prolonged decompression with subsequent lowering of the risk for PEP. Findings from two retrospective studies showed that longer PDS was more effective in reducing the risk of post-ERCP hyperamylasemia and the frequency of PEP compared with the shorter PDS. We conducted this trial to test whether 7cm PDS was superior to 5cm PDS in PEP prevention in high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

1. Un-intentional pancreatic duct cannulation:

   * 2 or more times;
   * 1 time with more than 10 minutes cannulation.
2. Double-wire technique;
3. High-risk patients:

met at least 1 of the major criteria

* Clinical suspicion of sphincter of Oddi dysfunction;
* Pancreatic sphincterotomy
* Delayed precut sphincterotomy
* ≥ 8 cannulation attempts
* Pneumatic dilatation of an intact biliary sphincter
* Ampullectomy

or met at least 2 or more of the minor criteria

* Age < 50;
* Female;
* Normal TBIL;
* ≥ 3 injections of contrast into the pancreatic duct with ≥ 1 injection to the tail of the pancreas;

Exclusion Criteria:

* Therapeutic PDS;
* Acute pancreatitis within 3 days;
* With a history of pancreatic surgery or biliary-enteric anastomosis;
* Pregnant or breastfeeding women;
* unwilling or inability to provide consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Post-ERCP Pancreatitis | 14 days
  The diagnosis of PEP was established if there was new onset of upper abdominal pain associated with an increased serum amylase level of at least 3 times the upper limit of normal range at 24 hours after the procedure, and hospitalization for at least 2 nights.

SECONDARY OUTCOMES:
Moderate to severe PEP | 14 days
  The severity classification of pancreatitis was defined according to the criteria of Cotton et al and the revised Atlanta criteria.
Other complications of ERCP | 14 days
  Other complications include post sphincterotomy bleeding, biliary infection, perforation, and any adverse outcomes possibly related to ERCP that required hospital admission or a prolonged hospital stay for further management.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi’an, Shanxi, China

REFERENCES:
- [Background] Domagk D, Oppong KW, Aabakken L, Czako L, Gyokeres T, Manes G, Meier P, Poley JW, Ponchon T, Tringali A, Bellisario C, Minozzi S, Senore C, Bennett C, Bretthauer M, Hassan C, Kaminski MF, Dinis-Ribeiro M, Rees CJ, Spada C, Valori R, Bisschops R, Rutter MD. Performance measures for ERCP and endoscopic ultrasound: a European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative. Endoscopy. 2018 Nov;50(11):1116-1127. doi: 10.1055/a-0749-8767. Epub 2018 Oct 19. PMID 30340220
- [Background] Sugimoto M, Takagi T, Suzuki R, Konno N, Asama H, Sato Y, Irie H, Watanabe K, Nakamura J, Kikuchi H, Waragai Y, Takasumi M, Hikichi T, Ohira H. Pancreatic stents for the prevention of post-endoscopic retrograde cholangiopancreatography pancreatitis should be inserted up to the pancreatic body or tail. World J Gastroenterol. 2018 Jun 14;24(22):2392-2399. doi: 10.3748/wjg.v24.i22.2392. PMID 29904246
- [Background] Olsson G, Lubbe J, Arnelo U, Jonas E, Tornqvist B, Lundell L, Enochsson L. The impact of prophylactic pancreatic stenting on post-ERCP pancreatitis: A nationwide, register-based study. United European Gastroenterol J. 2017 Feb;5(1):111-118. doi: 10.1177/2050640616645434. Epub 2016 Jul 8. PMID 28405329